CLINICAL TRIAL: NCT07364175
Title: Standard of Care or Weight Loss Drug Therapy in Obesity-related Hypertension - Pilot Study
Brief Title: A Trial Within Cohort Feasibility Study Design Comparing Standard of Care Versus Weight Loss (Achieved Through Tirzepatide) for Obesity-related Hypertension in Young Adults
Acronym: SOLUTION-Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, James Goodman, Consultant Physician and Clinical Pharmacologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R+D: A097457, REC: 25/WA/0268
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Obesity & Overweight
Keywords: hypertension; obesity; overweight; tirzepatide; GLP-1
MeSH Terms: conditions — Hypertension; Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: The study will utilise a modified trial within cohort (TwiC) design for patients under the hypertension/clinical pharmacology clinic. Those who meet the eligibility criteria for randomisation will be randomised to being approached for either:
  (i) 6 months of treatment with a combined GLP-1/GIP receptor agonist, Tirzepatide [Group A - Weight loss arm] (ii) Standard anti-hypertensive treatment and attendance at a 6-month combined research/clinical follow-up visit [Group B - Standard of Care (SoC) arm].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirzepatide [weight loss arm] (Experimental): 6 months of treatment with a combined GLP-1/GIP receptor agonist, tirzepatide
  Interventions: Drug: Tirzepatide
- Lifestyle advice and anti-hypertensive medications [standard of Care arm] (Active Comparator)
  Interventions: Drug: Anti-Hypertensive medications

INTERVENTIONS:
Drug: Tirzepatide — 2.5mg for 4 weeks, 5mg for 4 weeks, 7.5mg for 4 weeks, 10mg for 12 weeks
  Arms: Tirzepatide [weight loss arm]
Drug: Anti-Hypertensive medications — Anti-hypertensive drug therapy as per local and national guidelines
  Arms: Lifestyle advice and anti-hypertensive medications [standard of Care arm]

SUMMARY:
Hypertension is the leading risk factor for death globally, affecting approximately 30% of adults in the United Kingdom. Obesity is also a serious and ongoing epidemic, with global obesity rates having more than tripled in men and doubled in women, since 1975. In the United Kingdom, 64% of the adult population are overweight or obese. Hypertension and obesity share a well-established association, with obesity being responsible for the development of hypertension in 40-78% of cases. In young adults, this link between body size and blood pressure (BP) is much stronger that in older adults. Since overweight and obesity are among the most common and modifiable causes of high BP, weight loss induced by lifestyle-changes is recommended for overweight or obese patients with hypertension. However, lifestyle interventions, even when successful, result in only moderate weight loss, which is not maintained in the majority of cases. A meta-analysis of randomised controlled trials demonstrated that lifestyle-interventions lead to an average net weight reduction of 5.1 kg, accompanied by a significant, but modest, ~4 mmHg reduction in BP. Weight loss interventions could play a crucial role in the treatment of obesity-related hypertension in young adults.

Glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) receptor agonists, originally developed for the treatment of type 2 diabetes, are safe and clinically effective anti-obesity drugs. Recent data show a 10-20% placebo-adjusted reduction in body weight in overweight or obese adults without diabetes using the GLP-1 analogue semaglutide or the dual GLP-1/GIP receptor agonist tirzepatide, with the majority of weight loss achieved within the initial six months. The substantial weight loss induced by these drugs is accompanied by a significant reduction in BP. Two recent meta-analyses showed that semaglutide is associated with a ~5 mmHg placebo-adjusted reduction in clinic systolic BP (SBP). A sub-study of the SURMOUNT-1 trial reported a ~10 mmHg reduction in 24-h ambulatory SBP with tirzepatide. Most participants in these studies were normotensive or had well-controlled hypertension. Furthermore, antihypertensive medication use declined amongst those receiving anti-obesity drugs meaning the BP-lowering effect of weight loss, elicited by these drugs, is probably underestimated. These data suggest that the new anti-obesity drugs could be effective in managing overweight or obesity-related hypertension. Furthermore, it may be possible to cure hypertension in at least some young adults, removing the need for life-long antihypertensive treatment. However, the magnitude and time course of BP reduction elicited by these new anti-obesity drugs remain uncertain.

The primary aim of this feasibility study is to assess the extent and trajectory of BP reduction achieved through intensive weight loss in overweight or obese adults with stage 1 hypertension and compare this to current standard of care measures which uses anti-hypertensive medications and lifestyle advice. The study will utilise a modified trial within cohort approach, using patients based within the clinical pharmacology/hypertension service at Addenbrooke's Hospital, Cambridge.

ELIGIBILITY:
Eligibility criteria for randomisation

Inclusion Criteria:

* Aged 18 to 40 years (inclusive)
* Body mass index (BMI) ≥27 kg/m2
* Clinical diagnosis of primary (essential) hypertension as per NICE guidance
* Unattended brachial SBP ≥135 and/or DBP ≥85 mmHg and <160/100 mmHg
* Maximum of one antihypertensive medication

Exclusion Criteria:

• Anything in medical notes suggesting unsuitable in the opinion of the investigator

Eligibility criteria for participation in weight loss arm

Inclusion criteria:

* Written informed consent
* Aged 18 to 40 years (inclusive)
* Body mass index ≥27 kg/m2
* Clinical diagnosis of primary (essential) hypertension as per NICE guidance
* Unattended brachial SBP ≥135 and/or DBP ≥85 mmHg and <160/100 mmHg
* Maximum of one antihypertensive medication

Exclusion criteria:

The presence of any of the following will preclude participant inclusion:

* Known or suspected secondary hypertension
* Hypersensitivity to any of the study drugs or excipients
* Currently taking drugs likely to have interactions with tirzepatide
* Diagnosis of type 1 or type 2 diabetes mellitus or current usage of insulin or other injectable drugs for the treatment of diabetes such as but not limited to GLP-1 and GIP receptor agonists
* Prior or planned surgical, endoscopic and/or device-based therapy treatment for obesity
* Self-reported, intentional or unintentional, change in body weight (over ~10%) within ~three months of screening
* Known heart failure or clinically significant valvular heart disease
* Implanted pacemaker or implantable cardioverter defibrillator (ICD)
* Second or third-degree AV block, sino-atrial block, sick sinus syndrome
* Known active malignancy including thyroid cancer
* Known renal impairment (creatinine >150µmol/L)
* Clinically significant neurological disease
* History of scleroderma
* Participants on anticoagulant therapy
* Known history of pancreatitis
* Known inflammatory bowel disease
* History of gallstones (unless previous cholecystectomy)
* Severe gastroparesis or gastric emptying abnormality
* Family history of multiple endocrine neoplasia
* Needle-phobia
* Planned pregnancy, current pregnancy, or breastfeeding
* Current involvement in the active treatment phase of other research studies
* Any other clinical reason which may preclude entry in the opinion of the investigator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Ambulatory systolic blood pressure | Baseline to week 24
  Change in daytime ambulatory systolic blood pressure in the weight loss arm

SECONDARY OUTCOMES:
Ambulatory diastolic blood pressure | Baseline to week 24
  Change in daytime ambulatory diastolic blood pressure in the weight loss arm
Clinic systolic blood pressure | Baseline to week 24
  Changes in clinic systolic blood pressure in the weight loss arm
Clinic diastolic blood pressure | Baseline to week 24
  Changes in clinic diastolic blood pressure in the weight loss arm
Clinic mean arterial pressure | Baseline to week 24
  Changes in clinic mean arterial pressure in the weight loss arm
Unattended systolic blood pressure | Baseline to week 24
  Changes in unattended systolic blood pressure in the weight loss arm
Unattended diastolic blood pressure | Baseline to week 24
  Changes in unattended diastolic blood pressure in the weight loss arm
Unattended mean arterial pressure | Baseline to week 24
  Changes in unattended mean arterial pressure in the weight loss arm
Body weight | Baseline to week 24
  Changes in body weight in the weight loss arm
Body fat | Baseline to week 24
  Changes in body fat in the weight loss arm
Waist:hip ratio | Baseline to week 24
  Changes in waist:hip ratio in the weight loss arm
Cardiac output | Baseline to week 24
  Changes in cardiac output in the weight loss arm
Peripheral vascular resistance | Baseline to week 24
  Changes in peripheral vascular resistance in the weight loss arm
Pulse wave analysis / pulse wave velocity | Baseline to week 24
  Changes in markers of pulse wave analysis and pulse wave velocity in the weight loss arm
Heart rate variability | Baseline to week 24
  Changes in heart rate variability in the weight loss arm
Renin | Baseline to week 24
  Changes in plasma renin in the weight loss arm
Aldosterone | Baseline to week 24
  Changes in plasma aldosterone in the weight loss arm
Plasma metanephrines | Baseline to week 24
  Changes in plasma metanephrines in the weight loss arm
Leptin | Baseline to week 24
  Changes in leptin in the weight loss arm
Insulin | Baseline to week 24
  Changes in plasma insulin in the weight loss arm
Lipid profile | Baseline to week 24
  Changes in the lipid profile in the weight loss arm
HbA1C | Baseline to week 24
  Changes in HbA1C in the weight loss arm
Estimated glomerular filtration rate | Baseline to week 24
  Changes in eGFR in the weight loss arm
N-terminal pro-B-type natriuretic peptide | Baseline to week 24
  Changes in NT-proBNP in the weight loss arm
Urine albumin:creatinine ratio | Baseline to week 24
  Change in urine albumin:creatinine ratio in the weight loss arm
24-hour urine sodium | Baseline to week 24
  Change in 24-hour urine sodium in the weight loss arm
24-hour urine aldosterone | Baseline to week 24
  Change in 24-hour urine aldosterone in the weight loss arm
Antihypertensive medications | Baseline to week 24
  Change in number of antihypertensive medications
Quality of life measures | Baseline to week 24
  Changes in quality of life questionnaire scores in the weight loss arm
Ambulatory systolic blood pressure | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in ambulatory sytolic blood pressure
Ambulatory diastolic blood pressure | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in ambulatory diastolic blood pressure
Clinic systolic blood pressure | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in clinic systolic blood pressure
Clinic diastolic blood pressure | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in clinic diastolic blood pressure
Clinic mean arterial pressure | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in clinic mean arterial pressure
Unattended systolic blood pressure | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in unattended systolic blood pressure
Unattended diastolic blood pressure | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in unattended diastolic blood pressure
Unattended mean arterial pressure | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in mean arterial pressure
Body weight | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group body weight
Body fat | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in body fat
Waist:hip ratio | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in waist:hip ratio
Cardiac output | At week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in cardiac output
Peripheral vascular resistance | At week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in peripheral vascular resistance
Pulse wave analysis / pulse wave velocity | At week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in markers of pulse wave analysis and pulse wave velocity
Heart rate variability | At week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in heart rate variability
Plasma renin | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in plasma renin
Plasma aldosterone | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in plasma aldosterone
Plasma metanephrines | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in plasma metanephrines
Lipid profile | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in lipid profile
HbA1C | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in HbA1C
Estimated glomerular filtration rate | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in eGFR
N-terminal pro-B-type natriuretic peptide | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in NT-proBNP
Urine albumin:creatinine ratio | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in urine albumin:creatinine ratio
24-hour urine sodium | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in 24-hour urine sodium
24-hour urine aldosterone | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in 24-hour urine aldosterone
Number of antihypertensive medications | Change from baseline to week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in the number of anti-hypertensive medications
Quality of life measures | At week 24 (weight loss arm) and 6 months (standard of care arm)
  Between-group comparison in quality of life questionnaire scores

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following publication, the data that support the findings of this study will be available from the Chief Investigator/corresponding author upon reasonable request
Supporting Information: Study Protocol, CSR
Access Criteria: Following publication, the data that support the findings of this study will be available from the Chief Investigator/corresponding author upon reasonable request